CLINICAL TRIAL: NCT04953520
Title: Ultrasound-CT Fusion Image-guided Minimally Invasive Interventional Treatment of Lumbosacral Nerve Roots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2017318
Record Dates: First submitted 2021-06-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-CT fusion imaging guidance (Experimental): The patient undergoes lumbar nerve root block guided puncture needle placement under the guidance of ultrasound-CT fusion imaging
  Interventions: Procedure: ultrasound-CT fusion imaging
- Pure ultrasound guidance (Active Comparator): The patient undergoes lumbar nerve root block guided puncture needle placement under the guidance of pure ultrasound guidance
  Interventions: Procedure: pure ultrasound guidance

INTERVENTIONS:
Procedure: ultrasound-CT fusion imaging — The patient undergoes lumbar nerve root block guided puncture needle placement under the guidance of ultrasound-CT fusion imaging
  Arms: Ultrasound-CT fusion imaging guidance
Procedure: pure ultrasound guidance — The patient undergoes lumbar nerve root block guided puncture needle placement under the guidance of pure ultrasound guidance
  Arms: Pure ultrasound guidance

SUMMARY:
The study is aimed at patients with low back and leg pain. The patients in the experimental group were guided by ultrasound-CT fusion imaging to insert the lumbar nerve root puncture needle.

Patients in the control group underwent the insertion of the lumbar nerve root puncture needle under the guidance of ultrasound alone.

DETAILED DESCRIPTION:
A total of 80 patients with low back and leg pain were randomly divided into two groups, 30 people in each group. The patients in the experimental group were guided by ultrasound-CT fusion imaging to insert the lumbar nerve root puncture needle.Patients in the control group underwent the insertion of the lumbar nerve root puncture needle under the guidance of ultrasound alone.Follow-up of VAS pain score after lumbar nerve root block treatment. This study aims to establish a standardized operation method and process for lumbosacral nerve ultrasound-CT fusion guided interventional pain treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who need lumbar nerve root block treatment

Exclusion Criteria:

1. Tumor patients
2. Patients who have had lumbar spine surgery before

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
1 month VAS pain score | VAS pain scores were performed 1 month after surgery
  Patients undergo VAS pain score after the sonographer performs selective lumbar nerve root block puncture
3 month VAS pain score | VAS pain scores were performed 3 month after surgery
  Patients undergo VAS pain score after the sonographer performs selective
6 month VAS pain score | VAS pain scores were performed 6 month after surgery
  Patients undergo VAS pain score after the sonographer performs selective

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Cui, Study Chair — Peking University Third Hospital
Locations (1):
- Department of Ultrasound Diagnosis, Peking University Third Hospital, Beijing, Beijing Municipality, China